CLINICAL TRIAL: NCT03316820
Title: A Randomized, Open Label, Four Period, Four Sequence, Single Dose, Crossover Study to Evaluate Relative Bioavailability of K0706 24 mg Tablet Formulation Relative to 24 mg Capsule Formulation Under Fasted Conditions and to Evaluate the Food Effect for Tablet Formulation in Healthy Subjects
Brief Title: Bioavailability Study of K0706 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLR_17_07
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): K0706 tablet
  Interventions: Drug: K0706
- Treatment B (Experimental): K0706 tablet
  Interventions: Drug: K0706
- Treatment C (Experimental): K0706 tablet
  Interventions: Drug: K0706
- Treatment D (Experimental): K0706 capsule
  Interventions: Drug: K0706

INTERVENTIONS:
Drug: K0706 — Study treatment with water after an overnight fast
Drug: K0706 — Study treatment with water after food

SUMMARY:
This is single-center, single-dose, randomized, open-label, four-period, four sequence crossover study to evaluate the relative bioavailability of K0706 24 mg tablet formulation relative to 24 mg capsule formulation under fasted conditions and to evaluate the food-effect for tablet formulation in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide written, informed consent for participation in the study in the compliance with the protocol requirements
2. Adult males or females aged between 18 and 55 years
3. Medically healthy on the basis of medical history and physical examination
4. Woman of childbearing potential must practice an acceptable method of birth control

Exclusion Criteria:

1. History of any major surgical or medical conditions within 4 weeks prior to dosing
2. History of blood transfusion and / or plasmapheresis within 4 weeks prior to dosing
3. Inability to swallow oral medication and / or difficulty to find peripheral access to veins or inability to undergo venipuncture
4. Any malignancy within the past 3 years (except for non-melanoma skin cancer or cervical cancer in situ)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-28 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
Observed peak plasma concentration | 72 hours

SECONDARY OUTCOMES:
Adverse event | 26 days

CONTACTS AND LOCATIONS:
Locations (1):
- SPARC Site 1, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No